CLINICAL TRIAL: NCT01367574
Title: A Phase II Double-Blind, Randomized, Parallel Group, Dose Ranging Study of Subcutaneous Methylnaltrexone in Patients With Opioid-Induced Bowel Dysfunction
Brief Title: Methylnaltrexone in Patients With Opioid-Induced Bowel Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, M.D., Progenics Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 251
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Bowel Dysfunction
Keywords: Opioid-induced bowel dysfunction
MeSH Terms: conditions — Intestinal Diseases; Opioid-Induced Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: SC MNTX
- Arm 2 (Experimental)
  Interventions: Drug: SC MNTX
- Arm 3 (Experimental)
  Interventions: Drug: SC MNTX

INTERVENTIONS:
Drug: SC MNTX — Dose 1
  Arms: Arm 1
Drug: SC MNTX — Dose 2
  Arms: Arm 2
Drug: SC MNTX — Dose 3
  Arms: Arm 3

SUMMARY:
This is a double-blind, randomized, parallel group, dose ranging study of subcutaneous methylnaltrexone to be conducted in patients with advanced medical illness and poorly controlled opioid induced constipation. Patients will be randomized to one of three fixed dose levels of SC MNTX.

ELIGIBILITY:
Inclusion Criteria:

1. Must have advanced medical illness (cancer, HIV, etc) and be receiving palliative care
2. Must be on opioid medication for at least 2 weeks with no expectation of significant change in regimen
3. Must have constipation
4. Must be 18 yrs or older

Exclusion Criteria:

1. Concurrent use of medications other than opioids which might interfere with gastrointestinal motility
2. Patients who received any experimental drug in the last 30 days
3. Patients with active peritoneal cancer (ovarian, etc.)
4. Patients with active diverticulitis or diverticulosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2002-04; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects who have a bowel movement within four hours of dosing | Up to 4 weeks
  To access the efficacy of various fixed unit doses of MNTX SC in patients with advanced medical illnesses and poorly controlled opioid-induced constipation.

SECONDARY OUTCOMES:
Number of subject with Adverse Events | Up to 4 weeks
  To access the tolerability of various fixed unit doses of MNTX SC in patients with advanced medical illnesses and poorly controlled opioid-induced constipation.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States